CLINICAL TRIAL: NCT06732596
Title: Sustaining Recovery for People on Opioid Agonist Treatment With Conversational Agents
Acronym: SARA RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-45380; 1R34DA058124-01A1 (NIH)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: Embodied conversational agent (ECA); Buprenorphine treatment; Medication for opioid use disorder (MOUD); Office Based Addiction Treatment; Supportive Application for Recovery Assistance (SARA); Smartphone delivered intervention
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups: 50 will receive the ECA intervention (including technical support, text message reminders, and monetary incentives) in addition to usual care, while 50 will receive only usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECA, technical support, additional ECA messages, and incentives (Experimental): Participants randomized into the intervention arm will be engaged in ECA use, technical support, additional ECA messages reminding the use of the ECA app on behalf of OBAT clinical staff, and monetary incentives.
  Interventions: Other: Embodied conversational agent (ECA); Other: Technical support; Other: Additional ECA messages; Other: Additional incentives
- Treatment as usual group (No Intervention): Participants randomized into this arm will receive treatment as usual

INTERVENTIONS:
Other: Embodied conversational agent (ECA) — The app with the ECA will be provided.
  Arms: ECA, technical support, additional ECA messages, and incentives
Other: Technical support — Technical support will include assistance downloading and setting up the app on the participant's phone, walking them through a brief demonstration, and answering any questions the participant has about how to use the app.
  Arms: ECA, technical support, additional ECA messages, and incentives
Other: Additional ECA messages — Weekly text messages will be provided reminding participants to use the app on behalf of OBAT clinical staff.
  Arms: ECA, technical support, additional ECA messages, and incentives
Other: Additional incentives — Additional incentives will be provided after logging into the app for 20 days followed by monthly lotteries for those who log in 15 days per month
  Arms: ECA, technical support, additional ECA messages, and incentives

SUMMARY:
This study aims to improve retention in buprenorphine treatment, a medication used for opioid use disorder, through the use of a smartphone-delivered recovery support intervention. The intervention involves an Embodied Conversational Agent (ECA), a virtual, animated computer agent designed to simulate natural face-to-face conversations. ECAs have been shown to help individuals manage their healthcare in other settings, and this study seeks to evaluate their potential in supporting patients on medication for opioid use disorder (MOUD).

DETAILED DESCRIPTION:
One hundred participants will be enrolled in the study from the Office-Based Addiction Treatment (OBAT) clinic at Boston Medical Center (BMC). The participants will be randomly assigned to one of two groups. In the intervention group, participants will engage in ECA use and will receive (1) technical support, (2) text message reminders, and (3) monetary incentives. Alternatively, participants will be randomized to the treatment as usual group where they do not access the ECA application. Assessments will be conducted in person at baseline and over the phone at 6 months and 12 months. At 3 and 9 months, research staff will make brief telephone contacts to confirm or update participant contact information. The primary outcome is retention in buprenorphine treatment over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Opioid Use Disorder (OUD)
* Within 30 days of intake at recruitment site (BMC OBAT)
* Possession of a smartphone that has minimum requirements
* English-speaking and reading
* Willing to release electronic health record (EHR) data
* Able to provide at least two alternate contacts who usually know how to get in touch with them
* Currently prescribed buprenorphine from an outpatient clinic

Exclusion Criteria:

* Incarceration anticipated within 12 months of enrollment
* Inability to comprehend the study protocol, defined as failing three times to answer correctly a set of questions during the consent process
* Inability to use the ECA app (i.e., due to markedly limited visual or auditory acuity or motor function required to interact with the ECA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants that stay engaged in buprenorphine treatment | 12 months
  Engaged in buprenorphine treatment or treatment retention is defined as a participant's treatment period of at least 365 days, including those with multiple disengagement and reengagement periods, as long as any gap in active prescriptions or receipt of injections is less than 60 days.

SECONDARY OUTCOMES:
Treatment retention at 6 months | 6 months
  Treatment retention is defined as a participant's treatment period of at least 365 days, including those with multiple disengagement and reengagement periods, as long as any gap in active prescriptions or receipt of injections is less than 60 days.
Treatment duration | 6 months. 12 months
  Treatment duration is defined as length of continuous buprenorphine treatment in days until first discontinuation and will be measured via electronic health record (EHR) prescription and injection data and supplemented with self-report. Discontinued buprenorphine treatment occurs once the EHR indicates that they haven't filled a buprenorphine prescription or haven't received a buprenorphine injection in the previous 60 days. The treatment discontinuation date will be the last day of an active prescription or injection received.
Opioid use | 6 months
  Opioid use will be measured by self-report via the modified Addiction Severity Index (ASI). The modified ASI is administered by the study staff for a list of 20 drugs/substances. For each the number of days of use and the route of administration of that drug/substance [0=N/A, 1=oral, 2=nasal, 3=smoking, 4=non-intravenous (IV), injection 5=IV, or 8=refused] is documented.
Changes in stigma based on the Substance Use Stigma Mechanism Scale (SU-SMS) | Baseline, 6 months
  The SU-SMS is a self reported, 18-item instrument. Each item has a 5 Likert frequency responses from 1=Never to 5=Very often. Total scores can range from 1 to 90 or from 1-30 for each of the three types of stigma [anticipated, enacted, and internalized]. Lower scores are correlated with less stigma.
Changes in stigma based on the Buprenorphine Treatment Stigma Mechanism Scale (BT-SMS) | Baseline, 6 months
  BT-SMS is a self reported, 25-item instrument. Each item has a 5 Likert frequency responses from 1=Never to 5=Very often. Total scores can range from 1 to 125 or from 1-45 for anticipated stigma, 1-45 for enacted stigma, and 1-35 for internalized stigma. Lower scores are correlated with less stigma.
Changes in recovery capital | Baseline, 6 months
  Changes in recovery capital will be measured by self-report via the Brief Assessment of Recovery Capital (BARC-10) which is a 10-item self administered instrument. Each item has 6 Likert possible responses where 1=Strongly disagree to 6=Strongly agree. Total scores can range from 1 to 60. Higher scores are correlated with more recovery capital.
Frequency of interaction with the ECA app | 6 months, 12 months
  Frequency of interactions with the ECA app will be collected via the app itself and provided to the BMC study team by the investigators at Northeastern University.
User attitude and satisfaction toward the ECA | 6 months
  User attitudes and satisfaction with the ECA app will be measured by self-report using the Bond subscale of the Working Alliance Inventory which is an investigator developed instrument. The Bond subscale has 6 questions with an analog type response from 'disagree completely' to 'agree completely'.

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Lunze, MD MPH DrPH, Principal Investigator — Boston Medical Center
Locations (1):
- Office-Based Addiction Treatment (OBAT) Clinic, BMC, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All data produced in the course of the project will be preserved and shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than at the time of publication. The duration of preservation and sharing of the data will be a minimum of 10 years after the end of the funding period.
Access Criteria: Data will be available by controlled access only. To access data users must submit an informal data request and signs BMC's Data Use Agreement (DUA), which limits subsequent use to the terms of the approved request and requires that users maintain data security, and refrain from any attempts to re-identify research participants or engage in any unauthorized uses of the data. To get access to the data, the user must submit a valid scientific question, include a statistical analysis plan. The MPIs will review the data request for scientific merit.